CLINICAL TRIAL: NCT06741579
Title: Mechanisms of Stimulation for Pain Alleviation
Acronym: M-SPA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Hah, Associate Professor of Anesthesiology, Perioperative and Pain Medicine (Adult Pain), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 76560; RM1NS128956-01A1 (NIH)
Record Dates: First submitted 2024-11-25; First posted 2024-12-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Neuropathic Pain in the Low Back and Legs; Peripheral Nerve Stimulation; Chronic Neuropathic Pain
Keywords: SPRINT PNS; NALU PNS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Conventional Medical Management (CMM) ONLY (Active Comparator)
  Interventions: Procedure: Conventional Care Regimen
- Peripheral Nerve Stimulation + Conventional Medical Management (PNS+CMM) (Experimental)
  Interventions: Device: Peripheral Nerve Stimulation; Procedure: Conventional Care Regimen

INTERVENTIONS:
Device: Peripheral Nerve Stimulation — This trial studies 2 FDA approved peripheral nerve stimulation devices that may reduce pain by sending electrical pulses to the nerve. The SPR SPRINT PNS System, a matchbox-sized, battery-powered wearable stimulator that uses a Mircrolead to deliver stimulation for pain relief. There is a small wireless hand-held remote that is used to activate/ adjust intensity of stimulation. Stimulation delivered by this device may interrupt pain signals and increase non-pain signals. The SPR SPRINT device is used for 60 days before the percutaneous Microlead(s) are removed. The Nalu PNS System, a dime-sized micro-implantable pulse generator (IPG) leveraging advanced microelectronics. The micro-IPG is powered by an externally worn therapy disc via radiofrequency worn over the IPG site with an adhesive clip applied to the skin or a relief belt. The device is remote-controlled by patients via an app.
  Arms: Peripheral Nerve Stimulation + Conventional Medical Management (PNS+CMM)
Procedure: Conventional Care Regimen — CMM-Only participants will receive conventional medical management for the duration of their time in the study.

SUMMARY:
This is a mechanistic randomized controlled trial of patients with chronic neuropathic pain (CNP) in the lower back, pelvis, and lower extremities, randomized to conventional medical management (CMM) or combined CMM and peripheral nerve stimulation therapy (PNS+CMM). Our goal is to compare treatment outcomes and trial response rate across the control and interventional device groups.

ELIGIBILITY:
Inclusion criteria for study participants

Adults aged 18 or older with clinically diagnosed unilateral CNP in the lower back, pelvis, or lower extremities, defined (per IASP classification) as persistent or recurrent neuropathic pain caused by a peripheral nerve lesion, history of a plausible nerve trauma, pain onset in temporal relation to the trauma, and pain distribution within the innervation territory of a peripheral nerve (or nerves).14 Negative and positive sensory symptoms or signs must be compatible with the innervation territory of the affected nerve. Can be post-traumatic, post-surgical, nerve compression, nerve ischemia, peripheral nerve injury, painful scar, nerve entrapment, mononeuropathy with or without loss of motor function

Patients enrolled in this study must already have been referred for or have an existing order for PNS therapy (either Nalu or SPR SPRINT), prior to consent and enrollment in this study, as part of their routine medical care. Patients cannot receive a referral for PNS device as part of the study procedures.

Positive response (at least 50% pain relief) to diagnostic nerve block(s) at the suspected site(s) of CNP.

Chronic (at least 6 months duration), intractable peripheral neuropathic pain; any nociceptive pain must be less prominent than the neuropathic pian.

Fluent in English writing, reading, and speaking

Ability and willingness to complete online assessments

Williness to refrain from physical activity for at least 7 days post-lead placement.

Willingness to refrain from physical activity or exercise causing muscle and/or joint soreness for 48 hours prior to QST, illicit drugs (marijuana) for 12 hours, as-needed (PRN) pain medications (e.g., NSAIDs, acetaminophen, opioids) for 12 hours prior to QST, and alcohol and nicotine on the day of QST prior to testing*

Exclusion Criteria:

Conditions causing inability to complete assessments (education, cognitive ability, mental status, medical status)

Active cancer diagnosis, active malignant neoplasm (metastatic or local) or evidence of paraneoplastic syndrome

Painful polyneuropathy (e.g., metabolic, autoimmune, familial, infectious disease, environmental toxins, treatment with neurotoxic drug)

Chronic central neuropathic pain (e.g., spinal cord injury, brain injury, multiple sclerosis)

Peripheral vascular disease

Diabetic neuropathy

Another pain diagnosis affecting the CNP site that could interfere with study procedures, accurate reporting and/or could confound evaluation of study endpoints (e.g., post-herpetic neuralgia)

Other active implantable devices (e.g., implantable cardioverter defibrillator, spinal cord stimulator, dorsal root ganglion stimulator, sacral nerve stimulator, deep brain stimulator, intrathecal pump)

Pregnancy, breastfeeding, or planning to conceive

Systemic infection or local infection at the anticipated PNS implant site

Immunocompromised state

Coagulation disorder, bleeding diathesis, platelet dysfunction, active anticoagulation

Interventional procedure and/or surgery to treat CNP in the last 30 days (subjects should be enrolled 30 days after last procedure, for prior ablative treatment must be enrolled at least 3 months after last procedure)

Untreated substance use disorder

Participating in another clinical trial with an active treatment arm

Numbness or loss of sensation at the bilateral thumbnails, peripheral neuropathy in the hands, circulatory or sensory problem in the hands*

Participants with a history of Raynaud's Syndrome*

Participants with SBP ≥150 and/or DBP ≥100*

*QST Inclusion/Exclusion Criteria. Participants can still be enrolled iif they have the QST-only exclusionary criteria have the QST-only exclusionary criteria, but QST will be modified based on responses

Additional Exclusion Criteria for Subjects receiving PET/MRI and PET/CT imaging at Stanford:

Prior radiation exposure of >2 rem total within the last 12 months

Standard contraindications that would preclude MRI including pacemakers or other electronic implants, metal foreign objects or fragments in the eye or body, and aneurysm clips.

Claustrophobia

Inability to understand and communicate with the investigators to complete the study related questionnaires

Females with positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Response: defined as 50% relief of average pain intensity at the area of lower back, pelvic, or lower extremity CNP. We will compare the means of a three-day diary of numeric rating scale of pain (NRS) intensity scores (0-10 scale) | Baseline to Month 3
  We will compare the mean of a three-day diary of numeric rating scale of pain (NRS) intensity scores (0-10 scale) at baseline to the mean of a three-day diary of NRS scores at 3 months comparing all participants randomized to CMM vs. PNS+CMM.

SECONDARY OUTCOMES:
Trial Response Rate | Baseline to 15 days
  Defined as 50% relief of average pain intensity comparing the mean of a three-day diary of NRS scores at baseline to the mean of a three-day diary of NRS scores at 15 days comparing participants randomized to CMM vs. PNS+CMM. This outcome will be assessed either 15 days after baseline assessments among participants randomized to CMM, 15 days after Nalu PNS trial lead placement, or 15 days after SPR Sprint PNS microlead placement.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hah, MD, MS., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- See also: SPR Therapeutics - SPRINT PNS System Overview — https://www.sprpainrelief.com/hcp/sprint-pns-system
- See also: NALU Neurostimulation - NALU PNS System Overview — https://nalumed.com/patients/peripheral-nerve-stimulator/